CLINICAL TRIAL: NCT04365010
Title: Effects of Low-chlorine Vs High-chlorine Crystalloid Solutions in Septic Shock Adults
Brief Title: Low-chlorine Vs High-chlorine Crystalloids in Septic Shock Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Ph.D, Southeast University, China
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RIN013-C
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Septic Shock
Keywords: crystalloids, septic shock, MAKE30
MeSH Terms: conditions — Shock, Septic | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective cluster-randomized, multiple-crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Bicarbonate Ringer's Injection (Experimental): 1. administration route and dosage：Intravenous infusion, 500~1000 ml/time. The dosage can be increased or decreased according to the age, weight and symptoms.
  2. rate: according to the the routine rate of fluid resuscitation of septic shock in the ICUs of Zhongda Hospital, School of Medicine, Southeast University.
  Interventions: Drug: Sodium Bicarbonate Ringer's Injection
- 0.9% Sodium Chloride Injection (Active Comparator): 1. administration route and dosage：Intravenous infusion, 500~1000 ml/time. The dosage can be increased or decreased according to the age, weight and symptoms.
  2. rate: according to the the routine rate of fluid resuscitation of septic shock in the ICUs of Zhongda Hospital, School of Medicine, Southeast University.
  Interventions: Drug: 0.9% Sodium Chloride Injection

INTERVENTIONS:
Drug: Sodium Bicarbonate Ringer's Injection — For each month of the trial, participating ICUs were assigned to use either Sodium Bicarbonate Ringer's Injection or 0.9% Saline for any intravenous administration of isotonic crystalloid. ICUs were randomly assigned to use Sodium Bicarbonate Ringer's Injection during even-numbered months and 0.9% Saline during odd-numbered months, or vice versa.
  Arms: Sodium Bicarbonate Ringer's Injection
Drug: 0.9% Sodium Chloride Injection — For each month of the trial, participating ICUs were assigned to use either Sodium Bicarbonate Ringer's Injection or 0.9% Saline for any intravenous administration of isotonic crystalloid. ICUs were randomly assigned to use Sodium Bicarbonate Ringer's Injection during even-numbered months and 0.9% Saline during odd-numbered months, or vice versa.
  Arms: 0.9% Sodium Chloride Injection

SUMMARY:
Fluid resuscitation is an important treatment in septic shock patients, however whether crystalloid composition affects septic shock patients outcomes remains unclear. According to previous studies, low-chlorine crystalloids could significantly reduce the incidence of kidney injury and 30-day mortality compared with high-chlorine crystalloids in critically ill adults. Therefore, we hypothesized that the use of low-chlorine crystalloids would result in a lower incidence of major adverse kidney events within 30 days (MAKE 30: overall incidence of death, new renal-replacement therapy, and persistent renal dysfunction) than high-chlorine crystalloids in septic shock adults.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old <age ≤ 85 years old;
2. Diagnosis of septic shock within 24 hours (sepsis 3.0);
3. Needing fluid resuscitation judged by clinicians;
4. The patient or the patient's legally acceptable representative signs the informed consent (signs within 24h of enrollment)

Exclusion Criteria:

1. Pregnant or lactating period;
2. Renal replacement therapy has been received or expected to receive within 6 hours;
3. Those who were previously enrolled in the study;
4. Estimated death within 24 hours;
5. Other situations that not suitable for enrollment judged by researchers.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
the composite of death and new receipt of renal-replacement therapy MAKE30 | up to 30 days
  overall incidence of death, new renal-replacement therapy, and persistent renal dysfunction within 30 days

IPD SHARING:
Plan to Share IPD: Undecided